CLINICAL TRIAL: NCT06375239
Title: Observational, Non-Interventional Study to Determine the Operational Feasibility and Measurement Properties of Endpoints in Patients with Retinal Degeneration
Brief Title: Observational Study to Assess Endpoint Operational Feasibility & Measurement Properties in Patients with Retinal Degeneration
Status: Recruiting | Type: Observational
Sponsor: Ray Therapeutics, Inc. (Industry)
Collaborators: The Vision Research and Assessment Institute (VRAI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RTx-VRAI-NHS01
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Retinitis Pigmentosa; Choroideremia; Stargardt Macular Dystrophy; Stargardt Disease; Geographic Atrophy from Age-related Macular Degeneration; X-lined Retinoschisis; Retinal Dystrophies
MeSH Terms: conditions — Retinitis Pigmentosa; Choroideremia; Stargardt Disease; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Retinitis Pigmentosa: Up to 40 patients with Retinitis Pigmentosa
- Choroideremia: Up to 40 patients with Choroideremia
- Stargardt Macular Dystrophy (Stargardt Disease): Up to 40 patients with Stargardt Macular Dystrophy also known as Stargardt Disease
- Geographic Atrophy from Age-related Macular Degeneration: Up to 40 patients with Geographic Atrophy from Age-related Macular Degeneration
- X-linked Retinoschisis: Up to 40 patients with X-linked Retinoschisis
- Other Retinal Dystrophies: Up to 40 patients with other retinal dystrophies

SUMMARY:
The Vision Research and Assessment Institute (VRAI) was established with the purpose of serving as a testing facility for efficacy endpoints for patients with Low Vision.

The mission of the VRAI is to enable the highest quality, standardized efficacy testing of patients with visual impairment.

The VRAI facilitates the development and refinement of existing endpoints specifically for testing patients with Low Vision.

DETAILED DESCRIPTION:
The VRAI is a state-of-the-art research institute specifically for patients with low or very low vision due to diseases of the retina of the eye. The Institute is staffed by highly experienced Low Vision specialists and provides a comfortable, familiar environment for patient testing.

The study is a non-interventional prospective cohort study of up to 40 patients for each disease condition (Retinitis Pigmentosa, Choroideremia, Stargardt Macular Dystrophy, Geographic Atrophy from Age-related Macular Degeneration, X-linked Retinoschisis or other retinal dystrophies ).

Patients are scheduled for an initial visit where they are tested on a series of efficacy tests. Thereafter, patients will be invited to attend for a further visit up to two weeks and then periodically for up to one year. The objectives of the study are to evaluate how well patients use their vision, how the tests relate to activities of daily living, establish clinical meaningfulness, assess the impact of disease progression and the precision and accuracy of each test in the context of their eye condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral retinitis pigmentosa, choroideremia, Stargardt macular dystrophy, geographic atrophy from age-related macular degeneration, X-linked retinoschisis or other retinal dystrophies confirmed from previous eye examination records
* Best-corrected visual acuity between 20/70 and HM in at least one eye as tested with clinic-based visual acuity method
* Reasonably fluent in English

Exclusion Criteria:

* Cognitive impairment, memory loss or dementia sufficient in severity to preclude informed consent or in the opinion of the investigator would prevent satisfactory completion of some or all of the testing.
* Any circumstance that in the opinion of the investigator, would interfere with participation in, or compliance with the study protocol
* Current pregnancy as reported by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to profound vision impairment diagnosed with retinitis pigmentosa, choroideremia, or Stargardt macular dystrophy (also known as Stargardt disease), geographic atrophy from age-related macular degeneration, X-linked retinoschisis or other retinal dystrophies
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Operational feasibility of testing moderate to profound vision impaired patients with various retinal dystrophies on a battery of visual assessments | 3 months
  Determining how many patients in the visual range 20/70 - HM (depending upon indication) can perform specific tests of visual function with a measurable score.

SECONDARY OUTCOMES:
To quantify patient-based measurement properties of each test modality (for the purposes of endpoint qualification) | 2 years
  Test-retest reliability on the same visit or on two different testing sessions on different days including determination of significant learning effects or other scoring variables that impact variability.
To quantify assessor-based measurement properties of each test modality (for the purposes of endpoint qualification) | 2 years
  Intra- and inter-grader variability for scoring of tests by test graders/raters. Assessments incorporating independent graders/raters will be assessed for within session and across session scoring reliability to ensure consistent methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Research and Assessment Institute, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No